CLINICAL TRIAL: NCT04328025
Title: Peer-Delivered HIV Self-Testing, STI Self-Sampling and PrEP for Transgender Women in Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC REF 0304-2019
Record Dates: First submitted 2020-03-20; First posted 2020-03-31 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: HIV; Sexually Transmitted Infections; PrEP; Transgender Women
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Randomization in a 1:1 ratio to either monthly peer delivery of HIV self-testing, STI self-sampling and PrEP (intervention arm) or quarterly in-clinic HIV testing and PrEP prescription (control arm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-Delivered HIV Self-Testing, STI Self-Sampling and PrEP (Active Comparator): For TGW in the intervention arm, peers will deliver HIVST and PrEP medications monthly in between quarterly clinic visits. Quarterly clinic-based testing will confirm accuracy of self-tests and identify inaccurate test results. Additionally, peers will remind TGW to self-test before opening a new PrEP bottle. They will also distribute STI self-sampling kits to TGW for own use, and with regular partners as needed. They will present smart phone instructional videos showing trans women how to self-collect pharyngeal, rectal and urine specimens for Neisseria gonorrhoeae and Chlamydia trachomatis testing.
  Peers will: a) motivate ongoing adherence; b) promote repeat HIV testing; and c) support PrEP use as problems arise. Self-sampling for STIs will be performed monthly by participants (with questions answered by the peer or other study staff as needed).
  Interventions: Other: Peer-delivered HIV self-testing, STI self-sampling and PrEP
- Facility-Delivered Care (No Intervention): Participants will receive facility-based HIV counseling, PrEP prescriptions condoms, risk reduction counseling, and management of sexually transmitted infections as standard of care.

INTERVENTIONS:
Other: Peer-delivered HIV self-testing, STI self-sampling and PrEP — Peer delivery of combination HIV prevention interventions to transgender women.
  Arms: Peer-Delivered HIV Self-Testing, STI Self-Sampling and PrEP

SUMMARY:
Transgender women (TGW) are at high risk for HIV infection, and are an important, under-researched population in sub-Saharan Africa. Globally, HIV acquisition risk among TGW is 13 times higher than other adults aged 15-49 years. In Uganda, HIV prevalence among TGW is 22% compared to 5.9% in the general population. Encouraging use of self-controlled HIV prevention tools - specifically, HIV self-testing (HIVST), STI self-sampling (STISS) and antiretroviral pre-exposure prophylaxis (PrEP) - to those testing HIV negative could decrease HIV incidence among African TGW. This R34 application proposes formative research and a pilot trial to develop an HIV prevention intervention for African transgender women (TGW). The investigators will evaluate whether peer-delivered combination HIV prevention increases testing uptake and empowers effective prevention decision making in TGW. Peer-led interventions are effective in increasing HIV and STI testing among other hard-to-reach vulnerable populations with high HIV prevalence but low testing coverage and are recommended by the World Health Organization. Exploring peer-delivery approaches to increase coverage of combination HIV prevention interventions is key to addressing research gaps in HIV epidemic control. However, little is known about the effectiveness of peer-delivered combination HIV prevention (HIVST, STISS and PrEP) for African TGW, or the best way to deliver care to this population. Key knowledge gaps include: 1) whether peer delivery increases testing rates and status knowledge, 2) the role of peers in creating demand for repeat testing and PrEP, and 3) how to optimize peer delivery of combination HIV prevention (HIVST, STISS and PrEP). To address these questions, this proposal seeks to conduct formative research to inform implementation of peer-delivered combination HIV prevention for African TGW (Aim 1), implement a pilot cluster randomized trial to evaluate the feasibility, acceptability and preliminary effectiveness of peer delivered combination HIV prevention (Aim 2), and conduct in-depth interviews to explore how peer-delivery of HIVST, STISS and PrEP influences prevention choices among TGW and sexual partners (Aim 3). This will be the first clinical trial, to our knowledge, to evaluate HIV self-testing and STI self-sampling in HIV-uninfected TGW. Pilot data from TGW and their partners will provide unique perspectives to inform HIV prevention delivery. The proposed proof-of-concept evaluation is uniquely positioned to improve prevention uptake for African TGW - a high-risk, marginalized, and underserved population. Rigorous application of mixed methodologies will generate actionable data for policy and programs, and provide a strong foundation for scalable implementation of cutting edge combination HIV prevention interventions for African TGW. The local transgender community is involved in study design, planning and implementation. This project is supported by the Ugandan Ministry of Health.

DETAILED DESCRIPTION:
Transgender women (TGW) are at high risk for HIV infection, and are an important, under-researched population in sub-Saharan Africa. Globally, HIV acquisition risk among TGW is 13 times higher than other adults aged 15-49 years. In Uganda, HIV prevalence among TGW is 22% compared to 5.9% in the general population. Encouraging use of self-controlled HIV prevention tools - specifically, HIV self-testing (HIVST), STI self-sampling (STISS) and antiretroviral pre-exposure prophylaxis (PrEP) - among those testing HIV negative could decrease HIV incidence among African TGW and secondary transmission to their sexual partners. This study comprises formative research and a pilot trial to develop an HIV prevention intervention for African TGW. The investigators will evaluate whether peer-delivered combination HIV prevention increases testing uptake and empowers effective prevention decision making in TGW. Peer-led interventions are effective in increasing HIV and STI testing among other hard-to-reach vulnerable populations with high HIV prevalence but low testing coverage and are recommended by the World Health Organization (WHO). Exploring peer-delivery approaches to increase coverage of combination HIV prevention interventions is key to addressing research gaps in HIV epidemic control. However, little is known about the effectiveness of peer-delivered combination HIV prevention (HIVST, STISS and PrEP) for African TGW, or the best way to deliver care to this population. Key knowledge gaps include: 1) whether peer delivery increases testing rates and status knowledge, 2) the role of peers in creating demand for repeat testing and PrEP, and 3) how to optimize peer delivery of combination HIV prevention (HIVST, STISS and PrEP).

To address these questions, this protocol describes formative research to inform implementation of peer-delivered combination HIV prevention for African TGW, followed by implementation of a pilot cluster randomized trial to evaluate the feasibility, acceptability and preliminary effectiveness of peer delivered combination HIV prevention, and in-depth interviews to explore how peer-delivery of HIVST, STISS and PrEP influences prevention choices among TGW and sexual partners. This will be the first clinical trial, to our knowledge, to evaluate HIV self-testing and STI self-sampling in HIV-uninfected TGW.

Aim 1: Conduct formative research to inform implementation of peer-delivered combination HIV prevention for African TGW.

Approach: Using the Social Ecological framework, the investigators will conduct in-depth interviews with TG peers, healthcare providers, civil society members, and Ministry of Health officials to: a) explore barriers and likely facilitators of HIVST, STISS and PrEP; and b) assess feasibility of respondent-driven sampling (RDS), the recruitment strategy for Aim 2.

Hypothesis: Respondents will provide insights into the feasibility and acceptability of peer-delivered HIVST, STISS and PrEP, and RDS recruitment.

Aim 2: Evaluate the feasibility, acceptability and preliminary effectiveness of peer-delivered combination HIV prevention (HIVST, STISS and PrEP) for African TGW by implementing a pilot cluster randomized controlled trial.

Approach: To pilot-test the effectiveness of this peer-delivered combination HIV prevention intervention, 10 TGW peer groups (1 peer and 8 participants) will be randomized in a 1:1 ratio to either monthly peer delivery of HIVST, STISS and PrEP (intervention arm) or quarterly in-clinic HIV testing and PrEP prescription (control arm). All will enroll at clinic and initiate PrEP. In between quarterly clinic visits, trained peers will: a) deliver additional HIVST kits and PrEP refills; b) distribute STI self-sampling kits to TGW for own use and with regular partners; and c) use smart phone instructional videos showing TGW how to self-collect pharyngeal, rectal & urine specimens. The investigators will provide: i) free testing and treatment of Neisseria gonorrhoeae and Chlamydia trachomatis; and ii) peer-assisted partner notification services. Primary outcomes are intervention feasibility, acceptability & PrEP adherence.

Hypothesis: Peer delivery will be feasible and acceptable, with higher uptake of testing and PrEP compared with control arm.

Aim 3: Explore how peer-delivery of HIVST, STISS and PrEP influences prevention choices among TGW and sexual partners.

Approach: To clarify the process through which peer-delivery may influence prevention choices, the investigators will conduct in-depth interviews with participants and their partners to assess perceptions and experiences with peer-delivered HIV/STI services, status disclosure, partner notification, behavior change and PrEP use.

Hypothesis: Peer-delivered combination HIV prevention will empower TGW to engage in prevention services, facilitate partner testing and efficiently identify persons with undiagnosed HIV and/or STIs.

ELIGIBILITY:
Inclusion Criteria:

* Report male sex assigned at birth
* Age ≥18
* If 14-17 years, qualification as a mature or emancipated minor due to having a sexually transmitted infection or cater for own livelihood
* Report condom-less anal intercourse in the past 6 months
* Able and willing to provide written informed consent
* Possess a valid recruitment coupon
* HIV-uninfected based on negative HIV rapid tests at the enrollment visit
* Adequate renal function, defined by normal creatinine levels and estimated creatinine clearance ≥60 mL/min
* Not infected with hepatitis B virus, as determined by a negative hepatitis B surface antigen test

Exclusion Criteria:

* Currently enrolled in a biomedical HIV prevention study
* Any clinically significant or chronic medical condition that is considered progressive or in the opinion of the investigator would make the participant unsuitable for the study, including severe infections requiring treatment such as tuberculosis, alcohol or drug abuse, or mental illness which precludes provision of informed consent
* Not planning to remain in the geographic area for the duration of the study

Min Age: 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identify as transgender women
Enrollment: 82 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of peer-delivered prevention as measured by number of HIV and STI self-test kits delivered to intervention arm participants | 12 months
  Proportion of kits successfully delivered
Acceptability of peer-delivered prevention as measured by 5-point Likert scales and qualitative interviews | 12 months
  Proportion of intervention arm participants using HIV/STI self-test kits
PrEP effectiveness as measured by intracellular tenofovir diphosphate levels in dried blood spots | 12 months
  Comparison of PrEP effectiveness by randomization arm

SECONDARY OUTCOMES:
Sexual risk behavior as measured by frequency of self-reported unprotected sex | 12 months
  Comparison of unprotected sexual frequency by randomization arm
STI incidence as measured by GeneXpert Chlamydia and Gonorrhoeae PRC testing | 12 months
  Comparison of STI incidence by randomization arm
PrEP initiation as measured by pharmacy records | 12 months
  Proportion of participants initiating PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mujugira, PhD, Principal Investigator — Infectious Diseases Institute
Locations (1):
- Infectious Diseases Institute Kasangati, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mujugira A, Karungi B, Nakyanzi A, Bagaya M, Nsubuga R, Sebuliba T, Nampewo O, Naddunga F, Birungi JE, Sapiri O, Nyanzi KR, Bambia F, Muwonge T, Gandhi M, Haberer JE. Peer-Delivered HIV Self-Testing, Sexually Transmitted Infection Self-Sampling, and Pre-exposure Prophylaxis for Transgender Women in Uganda: A Randomized Trial. J Acquir Immune Defic Syndr. 2024 Oct 1;97(2):125-132. doi: 10.1097/QAI.0000000000003471. PMID 39250646
- [Derived] Mujugira A, Nakyanzi A, Nabaggala MS, Muwonge TR, Ssebuliba T, Bagaya M, Nampewo O, Sapiri O, Nyanzi KR, Bambia F, Nsubuga R, Serwadda DM, Ware NC, Baeten JM, Haberer JE. Effect of HIV Self-Testing on PrEP Adherence Among Gender-Diverse Sex Workers in Uganda: A Randomized Trial. J Acquir Immune Defic Syndr. 2022 Apr 1;89(4):381-389. doi: 10.1097/QAI.0000000000002895. PMID 34954718